CLINICAL TRIAL: NCT04232813
Title: Evaluation of the Acceptability and Efficacy of 10 Micrograms of Estradiol Vaginal Tablets vs Promestriene Vaginal Cream
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Palacios (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-AVV2019
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Vulvovaginal Atrophy
Keywords: Vaginal dryness; Vaginal soreness; Vaginal irritation; Dyspareunia
MeSH Terms: conditions — Dyspareunia | interventions — Estradiol; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Intervention Model Description: A Prospective, monocentric, open-label, randomized, parallel-group study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estradiol 10 micrograms vaginal tablets (Active Comparator): One tablet intravaginally once daily for two weeks. Thereafter one tablet twice per week with at least a 3-days interval between treatments to maintain therapeutic response.
  Interventions: Drug: Estradiol 10 MCG Vaginal Tablet [VAGIFEM]
- Promestriene 10mg./g vaginal cream (Active Comparator): One application once daily intravaginally for two weeks. Thereafter one application twice per week with at least a 3-days interval between treatments to maintain therapeutic response.
  Interventions: Drug: Promestriene Vaginal

INTERVENTIONS:
Drug: Estradiol 10 MCG Vaginal Tablet [VAGIFEM] — To insert the tablets the patient must use the applicator provided in the way explained in the prospectus.
  Arms: Estradiol 10 micrograms vaginal tablets
Drug: Promestriene Vaginal — To insert the cream the patient must use the applicator provided in the way explained in the prospectus.
  Arms: Promestriene 10mg./g vaginal cream

SUMMARY:
Evaluation of the Acceptability and Efficacy of 10 Micrograms of Estradiol Vaginal Tablets vs Promestriene Vaginal Cream in postmenopausal women aged 45 years or older, with one or more moderate to severe symptoms of vulvovaginal atrophy (dryness, dyspareunia, soreness or irritation).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 45 years or older. Women will be considered postmenopausal with more than 12 months since last menstrual period
* Women who have read and signed the Informed Consent Form
* Women with an intact uterus
* One or more vaginal symptoms (dryness, soreness, irritation, dyspareunia) rated as moderate to severe. Symptoms are moderate if the patient needs a treatment and feels discomfort. Symptoms are severe if the patient needs a treatment, and feels such a degree of discomfort that this could severely impact the subject's daily activities.
* Blood estradiol concentration of 30 pg/ml or less .

Exclusion Criteria:

* Women who have not signed the Informed consent Form
* Women who had a known or suspected history of breast carcinoma
* Estrogen dependent neoplasia. Women with a known, past or suspected Estrogen-dependent malignant tumours such as endometrial or ovarian cancer
* Positive or suspicious mammogram results
* Any systemic malignant disease
* Hormone therapy treatment (sex hormones or vaginal treatments or steroids) in the last three months
* Women who had abnormal vaginal bleeding or uterine bleeding of unknown cause
* Vaginal infection requiring treatment
* Previous or current venous thromboembolism (deep venous thrombosis, pulmonary embolism) Untreated endometrial hyperplasia Known thrombophilic disorders (e.g. protein C, protein S, or antithrombin deficiency) Active or previous arterial thromboembolic disease (e.g. angina, myocardial infarction) Acute liver disease, or history of liver disease as long as liver function tests have failed to return to normal Known Hypersensitivity to the active substances or to any of the excipients Porphyria
* Any serious disease or chronic condition that could interfere with study compliance
* History of thrombolytic disorders
* Use of vaginal contraceptives (DIU, vaginal ring…)
* Participation in another clinical trial in the last three months.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Vulvovaginal Symptoms | Change from Baseline, at week 4 and at week 12
  Percentage of patients with vulvovaginal atrophy that accept 17B-Estradiol vaginal tablets vs promestriene vaginal cream after 12 weeks

SECONDARY OUTCOMES:
Evaluation of relief of atrophic vaginitis symptoms using intensity ratings of none, mild, moderate or severe of dryness and dyspareunia. | Change from Baseline, at week 4 and at week 12
  Percentage of women that verify a relief of atrophic vaginitis dryness, dyspareunia, soreness and irritation symptoms in the questionnaires provided at Visit 1 and Visit 2 compared to intensity of those symptoms at screening visit.
Evaluation of changes in ph. | Change from Baseline, at week 4 and at week 12
  Percentage of women with changes in pH at Visit 1 and Visit 2 compared to Screening Visit. Comparison with the two groups
Evaluation of vaginal maturation index by Pap smear. | Change from Baseline, at week 4 and at week 12
  Percentage of woman with changes in vaginal maturation index by Pap smear at Visit 2 compared to Screening Pap smear and comparison between groups.
Evaluation of changes in soreness and irritation. | Change from Baseline, at week 4 and at week 12
  Percentage of women that verify a relief of atrophic vaginitis dryness, dyspareunia, soreness and irritation symptoms in the questionnaires provided at Visit 1 and Visit 2 compared to intensity of those symptoms at screening visit.
Occurrence of adverse events | Change from Baseline, at week 4 and at week 12
  Number of adverse events
Evaluation of endometrium thickness using vaginal ultrasound | Change from Baseline, at week 4 and at week 12
  Percentage of women with changes in endometrium thickness at Visit 2 compared to Screening Visit and comparison between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Palacios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palacios S, Ramirez M, Lilue M. Efficacy of low-dose vaginal 17beta-estradiol versus vaginal promestriene for vulvovaginal atrophy. Climacteric. 2022 Aug;25(4):383-387. doi: 10.1080/13697137.2021.1998436. Epub 2021 Nov 23. PMID 34813408